CLINICAL TRIAL: NCT04368130
Title: SIGNAL:Identifying Behavioral Anomalies Using Smartphones to Improve Cancer Care
Acronym: SIGNAL
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The anomaly detection system is still under development and is not ready to test.
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Alexi A. Wright, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-246; R21NR018532-02 (NIH)
Record Dates: First submitted 2020-04-27; First posted 2020-04-29 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Carcinoma; Uterine Cancer; Cervical Cancer; Gynecologic Cancer
Keywords: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Carcinoma; Uterine Cancer; Cervical Cancer; Gynecologic Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Uterine Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SIGNAL (Experimental): Program to explore the feasibility and acceptability of a smartphone-based real-time behavioral anomaly detection system (SIGNAL).
  Patients will download the adapted Beiwe app onto their smartphones for a 6-month period and investigators will collect passive smartphone sensor data and active PRO data bi-weekly.
  Interventions: Behavioral: SIGNAL

INTERVENTIONS:
Behavioral: SIGNAL — SIGNAL is a smartphone-based mobile health intervention designed to improve important outcomes in cancer patient patients (e.g., symptom burden, physical functioning).
  Patients will download the adapted Beiwe app for a 6-month period and investigators will collect passive smartphone sensor data and active PRO data bi-weekly.

SUMMARY:
This research study is testing the use of a smartphone app to identify clinically meaningful changes in the behaviors of patients' with gynecological cancers by using passively collected smartphone data.

DETAILED DESCRIPTION:
This is a pilot study of patients with advanced gynecologic cancers and oncology providers from the Dana-Farber Cancer Institute's Gynecologic Oncology Program to explore the feasibility and acceptability of a smartphone-based real-time behavioral anomaly detection system (SIGNAL).

The research study procedures include screening for eligibility and study interventions including smartphone data collection, surveys, and a brief interview once you have completed the study to learn more about your experiences on the study.

Participants will download the adapted Beiwe app for a 6-month period and the investigators will collect passive smartphone sensor data and active PRO data bi-weekly.

ELIGIBILITY:
Inclusion Criteria:

* Women >18 years of age with newly diagnosed ovarian cancer (i.e. prior to completion of cytoreductive surgery-whether primary or interval cytoreductive surgery).
* Own a smartphone (Android or iOS).
* Capable of downloading and running the study apps.
* Can read and provide informed consent in English.
* Do not have cognitive or visual impairments that would preclude use of the app.

Exclusion Criteria

* Patients will be ineligible if they are participating in an investigational drug treatment trial that requires structured symptom or toxicity reporting at the time of enrollment.
* Patients with severe cognitive impairments or who appear too weak, emotionally distraught, agitated or ill to participate, as judged by either the research study staff or an oncology provider, will be excluded.
* Patients who are unable to provide informed consent in English will be excluded because the smartphone app is only available in English at this time.
* Children and young adults up to age 17 will be excluded because the diagnosis of metastatic gynecologic cancers in this age group is rare and the proposed instruments are not designed for people of those ages.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Rate of enrollment | 6 Months
  Feasibility will be demonstrated if ≥50% of eligible participants enroll
Rate of completion | 6 Months
  Feasibility will be demonstrated if ≥50% of eligible participants adhere to the smartphone app
Burden rate | 6 Months
  Acceptability will be defined as: <30% of patients rate the study as burdensome.

CONTACTS AND LOCATIONS:
Overall Officials: Alexi A. Wright, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu